CLINICAL TRIAL: NCT00991198
Title: The Role of Topically Dissolved Oxygen (TDO) to Ameliorate Signs of Photodamage in Individuals With Multiple Skin Conditions A Double-Blind, Placebo Controlled Comparative Trial
Brief Title: The Role of Topically Dissolved Oxygen (TDO) to Ameliorate Signs of Photodamage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aria Aesthetics Inc. (Industry)
Responsible Party: Larry Rheins, PhD/President, Aria Aesthetics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFLOTDO002
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Rosacea; Acne Vulgaris; Atopic Dermatitis; Seborrheic Dermatitis
Keywords: Topically dissolved oxygen; inflammatory cutaneous disease; rosacea; acne vulgaris; atopic dermatitis; seborrheic dermatitis; photodamage
MeSH Terms: conditions — Rosacea; Acne Vulgaris; Dermatitis, Atopic; Dermatitis, Seborrheic | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Aria Regimens 0.5% conc
  Interventions: Drug: Topical oxygen
- B (Experimental): Aria Regimen (5 products) 0.25% conc
  Interventions: Drug: Topical oxygen
- C (Placebo Comparator): Aria Regimen Control without O2
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Topical oxygen — 0.5% concentration of Topical oxygen
  Arms: A
Drug: Topical oxygen — 0.25% concentration topical oxygen
  Arms: B
Drug: placebo — no O2
  Arms: C

SUMMARY:
This study is an evaluation of the role of topical dissolved oxygen to lessen visible signs of photodamage using a select regimen of topical dissolved oxygen containing cosmeceutical products. Evaluation of the overall skin tolerability of topical dissolved oxygen (safety) utilizing the regimen of products.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be female, 25-60 years old in good general health;
* Subjects must be Fitzpatrick Types I, II, III, IV, V
* Subjects must be willing to forgo the use of facial cosmetics (e.g. facial moisturizers,creams, foundations, blush, etc.) during the course of the study.
* Subjects may ONLY use facial regimen of products provided by sponsor(lipstick, lip gloss, and eye mascara permitted).

Exclusion Criteria:

* Known sensitivity to any of the test material ingredients.
* Routine high dosage use of anti-inflammatory medications (aspirin, ibuprofen, corticosteroids), immunosuppressive drugs or antihistamine medications (steroid nose drops and/or eye drops are permitted) (one-8lmg or 325mg aspirin okay) (birth control is okay but needs to be reported).
* Use of topical OTC/Rx drugs or other cosmetics at the test sites.
* Immunological disorders such as HIV positive and systemic lupus erythematosus (interview only)
* Participation in any clinical study within the last four weeks.
* Pregnant or lactating women (interview only).
* Damaged skin in or around test sites (including sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test site).

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
skin grading evaluation of photodamage | 8 weeks

SECONDARY OUTCOMES:
stratum corneum hydration (skin capacitance) | 8 weeks
bioinstrumental assessment of skin "melanin" lightening, and lesional erythematous sites | 8 weeks
bioinstrumental assessment of skin texture, scaliness (desquamation) | 8 weeks
punch biopsy histopathologic examination (H&E, and immunohistochemistry for Aquaporin 3, and Filaggrin) | 8 weeks
RT-PCR collagenase , and hypoxia-inducible factor-1 alpha | 8 weeks
product performance | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consultants Inc.
Locations (1):
- Dermatology Consultants Inc, High Point, North Carolina, United States